CLINICAL TRIAL: NCT03268629
Title: The Efficacy of a Mindfulness-Based Intervention for Insomnia ('Mindfulness-Based Joyful Sleep') in Young and Middle-aged Individuals With Insomnia in China: Study Protocol of a Randomized Controlled Trial
Brief Title: 'Mindfulness-Based Joyful Sleep' Intervention in Young and Middle-aged Individuals With Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Chen Pan, Principal Investigator, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-S236
Record Dates: First submitted 2017-08-27; First posted 2017-08-31 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Insomnia
Keywords: Insomnia; Mindfulness-based Intervention; Mindfulness Meditation; Tai Chi; Inflammation; NF-κB
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Joyful Sleep (Experimental): The proposed 'Joyful Sleep' program will be conducted weekly, 2 hours per session, 8 sessions, group-based in mindfulness. The content and skills are based upon MBSR, MAPs and Tai Chi. The proposed topics include: 1) mindfulness and insomnia, 2) mindful awareness of stress, 3) mindful working with thoughts, 4) mindful working with emotions, 5) mindful interactions, 6) moving mindfulness meditation: the first taste of Tai Chi, 7) moving mindfulness meditation: the second taste of Tai Chi, 8) dealing with obstacles of mindful practices and wrap-up. Mindfulness practices embedded in the program will include mindfulness breathing meditation, body scan meditation, sitting meditation, standing meditation, walking meditation, Taichi, and daily life meditation.
  Interventions: Behavioral: Mindfulness-Based Joyful Sleep
- CBT-I (Active Comparator): The CBT-I is a weekly, 2-hour, 8 session, group-based program. CBT-I includes 4 central components: stimulus control, sleep restriction, relaxation training and cognitive therapy. The aim of CBT-I is to reduce sleep-related physiologic and cognitive arousal so that restorative sleep function can be re-established.
  Interventions: Behavioral: CBT-I

INTERVENTIONS:
Behavioral: Mindfulness-Based Joyful Sleep — The proposed "Mindfulness-Based Joyful Sleep" program will be conducted weekly, 2 hours per session, 8 sessions, group-based program in mindfulness.
  Other Names: Mindfulness based intervention for insomnia
  Arms: Mindfulness-Based Joyful Sleep
Behavioral: CBT-I — The CBT-I program was delivered to groups of 10-15 individuals over the course of eight, weekly, 2-hour sessions, for a total of 16 contact hours.
  Arms: CBT-I

SUMMARY:
The primary objective of this proposed three-year (June 01, 2018 to May 31,2020) project is to verify the effect of 'Mindfulness Based Joyful Sleep' (MBJS) intervention on young and middle-aged individuals with insomnia in China and preliminarily explore inflammatory response for the intervention of insomnia applied by it. Previous researches show that Mindfulness-Based Interventions may relieve insomnia, it is hypothesized that MBJS will be an effective, feasible and affordable insomnia intervention program in China.

DETAILED DESCRIPTION:
Background：Insomnia is a public health problem attracting extensive attention. Due to the risks of side effect and drug dependence from the drug treatment of insomnia, the non-drug treatment has gradually drawn the attention of clinician. In recent years, Mindfulness-Based Interventions originating from the Eastern culture has created a trend in the application and research of psychological and physical health fields in western countries, and been found to be capable of effectively curing or alleviating many psychosomatic diseases and possibly results in the reversion of gene operation mode and the reduction of inflammation risk. Researches show that Mindfulness-Based Interventions may relieve insomnia, but existing research samples and strict randomized controlled trial are insufficient and its application mechanism is full of uncertainty. In China, empirical research strictly designed is even scarce in such field. At the earlier stage, investigators have designed a intervention scheme for insomnia intervention ('Mindfulness-Based Joyful Sleep') with mindfulness-based meditation and Tai Chi as core technology, and in combination with Chinese culture and have made preliminary application.

Objectives：This study is expected to verify the effect of 'Mindfulness-Based Joyful Sleep' program on young and middle-aged patients with insomnia in China and preliminarily explore the genetic level inflammation mechanism for the intervention of insomnia applied by it.

Methods: Investigators will conduct a 2-arm randomized controlled trial to evaluate the efficacy of mindfulness-based intervention for insomnia ('Mindfulness-Based Joyful sleep'). Patients with insomnia at the age of 18-59 in China will be recruited for this study.The two steps to be implemented include: 1) conducting a pilot study to finalize the design of 'Mindfulness-Based Joyful sleep'program and evaluate the feasibility, acceptability and preliminary outcomes of the'Mindfulness-Based Joyful sleep' program: The final sample is expected to include18 patients who meet inclusion criteria. Participants will receive 8-week 'Mindfulness-Based Joyful sleep' intervention. The efficacy of 'Mindfulness-Based Joyful sleep' program will be assessed by PSQI, and feasibility and acceptability of 'Joyful Sleep' program will be examined by attendance, completion of homework and feedback of participants on the feeling of the program collected by a focus group. 2) conducting a randomized controlled trial to evaluate the efficacy of ''Mindfulness-Based Joyful sleep'' program: The final sample is expected to include 70 patients who meet inclusion criteria. Participants will be randomly assigned to one of 2 groups, receiving'Mindfulness-Based Joyful sleep'intervention, or receiving 'Cognitive Behavior Therapy for insomnia (CBT-I)'. Participants will be assessed at 3 time points by PSG, Sleep Diary, self-reported measures including PSQI, ISI, CPSS, BDI, STAI and bio-indicator (NF-κB) at baseline, the end of the Intervention Period, and at a 3-month follow-up.

Implications: This proposed study has important implications in providing valuable insights into bridging the gap between need and services received for insomnia interventions in China. If the 'Mindfulness-Based Joyful Sleep' Intervention can be used effectively, it can also be popularized to many other patients with insomnia in China in future.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 59 years
2. Diagnosis of insomnia disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th ed (DSM-V)
3. Fully conscious
4. Junior high school or higher education degree
5. No language impairment or communication disorders
6. Willing to participate in the study

Exclusion Criteria:

1. Cognitive impairment
2. Somatic disorders, including but not limited to cardiovascular disease, cerebrovascular diseases, endocrine diseases, autoimmune diseases, and tumors
3. Mental disorders, including but not limited to schizophrenia, mood disorders, anxiety disorders, trauma and stress related disorders, substance related disorders
4. Pregnant or lactating women
5. Currently taking any prescribed medication
6. Currently participating in any mindfulness practice for 15 minutes per day (e.g. yoga, Tai Chi, qigong, meditation)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
change of sleep quality | Outcomes will be evaluated at baseline, the end of the 8-week Intervention Period, and at a 3-month follow-up
  Sleep quality will be measured with Pittsburgh Sleep Quality Index (PSQI)

SECONDARY OUTCOMES:
change of perceived stress | Outcomes will be evaluated at baseline, the end of the 8-week Intervention Period, and at a 3-month follow-up
  Perceived stress will be assessed by Perceived Stress Scale (PSS). The PSS has 14 items. Items are rated on a 5-point Likert-type scale, with higher total scores indicating higher perceived stress (0-13, low perceived stress; 14-26, moderate perceived stress; 27-40, high perceived stress).
change of anxiety | Outcomes will be evaluated at baseline, the end of the 8-week Intervention Period, and at a 3-month follow-up
  Anxiety will be assessed by State-Trait Anxiety Inventory (STAI). The STAI has 20 items for assessing trait anxiety (TAI) and 20 items for assessing state anxiety (SAI). All items are rated on a 4-point scale, with higher total scores indicate greater anxiety.
change of depression | Outcomes will be evaluated at baseline, the end of the 8-week Intervention Period, and at a 3-month follow-up
  Depression will be assessed by Beck Depression Inventory (BDI). The BDI consists of 21 items. All items are rated on a 4-point scale, with higher total scores indicating more severe depression (31-40 indicates severe depressive symptoms and scores > 40 indicate extreme depressive symptoms).
change of nuclear factor-κB (NF-κB) | Outcomes will be evaluated at baseline, the end of the 8-week Intervention Period, and at a 3-month follow-up
  NF-κB (nuclear factor-κB) is a collective name for inducible dimeric transcription factors composed of members of the Rel family of DNA-binding proteins that recognize a common sequence motif. NF-κB is found in essentially all cell types and is involved in activation of an exceptionally large number of genes in response to infections, inflammation, and other stressful situations requiring rapid reprogramming of gene expression. NF-κB is clearly one of the most important regulators of proinflammatory gene expression.
change of sleep quantity | Outcomes will be evaluated at baseline, the end of the 8-week Intervention Period, and at a 3-month follow-up
  sleep quantity will be measured with Polysomnography (PSG).
change of severity of Insomnia Symptoms (ISI) | Outcomes will be evaluated at baseline, the end of the 8-week Intervention Period, and at a 3-month follow-up
  Severity of Insomnia Symptoms will be measured with Insomnia Severity Index (ISI). The ISI comprises 7 items, which are each rated on a five-point scale. Total scores range from zero to 28. ISI clinical cut points are categorized as: no insomnia (zero to seven), subthreshold insomnia (eight to 14), moderate insomnia (15-21), and severe insomnia (22-28).

CONTACTS AND LOCATIONS:
Overall Officials: Pan Chen, M.D.，Ph.D., Principal Investigator — Central South University
Locations (1):
- Thrid Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
data of participants' assessment result on PSG, Sleep Diary, PSQI, ISS, CPSS, BDI, STAI, NF-κB during intervention will be shared with other researchers through published articles.
Supporting Information: Study Protocol
Time Frame: data will be made available within 6 months of study completion and no time limitation.
Access Criteria: the data will become available on the database which includes the journal publishing the study.

REFERENCES:
- [Derived] Pan C, Wang X, Deng Y, Li P, Liao Y, Ma X, Yang GP, Dai L, Tang Q. Efficacy of mindfulness-based intervention ('mindfulness-based joyful sleep') in young and middle-aged individuals with insomnia using a biomarker of inflammatory responses: a prospective protocol of a randomised controlled trial in China. BMJ Open. 2019 Jul 10;9(7):e027061. doi: 10.1136/bmjopen-2018-027061. PMID 31296508